CLINICAL TRIAL: NCT01435122
Title: A Phase II Study of Axitinib in Advanced Carcinoid Tumors
Brief Title: A Study of Axitinib in Advanced Carcinoid Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Comprehensive Cancer Network (Network); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-16692
Record Dates: First submitted 2011-09-14; First posted 2011-09-15 (Estimated); Results first posted 2017-05-25 (Actual); Last update posted 2018-10-02 (Actual); Status verified 2018-08

CONDITIONS: Carcinoid Tumor
Keywords: progressive advanced carcinoid tumors; advanced; unresectable; metastatic; cancerous tumors; neuroendocrine; digestive tract; lungs; renal; ovarian; thymic; hepatic
MeSH Terms: conditions — Carcinoid Tumor; Neoplasm Metastasis | interventions — Axitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Axitinib Administration (Experimental): The investigational drug used in this study is axitinib, and is available as tablets.
  You will take the tablet orally with food. Doses should be taken around 12 hours apart continuously, without scheduled breaks. If you vomit anytime after taking a dose do not take another tablet to "make up the dose" but instead continue taking your next dose as planned.
  Any missed dose may be taken late (up to 3 hours before the next scheduled dose); otherwise it should be skipped. If doses are missed or vomited, please keep track of this and report at your next visit.
  Interventions: Drug: Axitinib

INTERVENTIONS:
Drug: Axitinib — Axitinib Administration as outlined in Arm description
  Other Names: AG013736; selective inhibitor of receptor tyrosine kinases

SUMMARY:
The main purpose of this study is to see whether Axitinib will help prolong the time that the patient's carcinoid tumors remain stable, and to examine their treatment response through testing. Researchers also want to find out if Axitinib is safe and tolerable.

DETAILED DESCRIPTION:
This is a bi-institutional, prospective phase II, open-label study. The target population is comprised of adult patients with histologically confirmed unresectable or metastatic carcinoid tumors. Carcinoid tumors are defined as well to moderately differentiated neuroendocrine tumors of the digestive tract and lungs. Patients with metastatic carcinoid tumors of unknown primary as well as rare primaries (renal, ovarian, thymic, hepatic) will also be eligible. Patients will be drawn from two institutions Moffitt Cancer Center (MCC) and The University of California, San Francisco (UCSF).

ELIGIBILITY:
Inclusion Criteria:

* Locally unresectable or metastatic well-and moderately-differentiated (low- or intermediate- grade) neuroendocrine tumors of the aerodigestive tract (e.g. foregut, midgut, and hindgut) and unknown primary site as well as rare primary sites (renal, ovarian, thymic, hepatic); Otherwise known as typical or atypical carcinoid tumors
* Measurable disease by Response Evaluation Criteria In Solid Tumors (RECIST) Criteria
* Functional or nonfunctional tumors allowed
* Evidence of progressive disease within 12 months of study entry
* Adequate hepatic function: total bilirubin ≤1.5 x upper limit of normal (ULN)mg/dl; aspartic transaminase (AST) ≤2.5 x ULN (≤5 x ULN if attributable to liver metastases)
* Adequate renal function: serum creatinine ≤ 1.5 x ULN
* Adequate bone marrow function: absolute neutrophil count ≥ 1,500/mm³; platelets ≥75,000/mm³
* Prothrombin time (PT) and activated partial thromboplastin time (aPTT) levels ≤1.5 x ULN (unless patients receiving coumadin anticoagulation in which case a stable international normalization ration (INR) of 2-3 is required).
* Urine protein <2+proteinuria (or <2 g proteinuria /24 hr)
* Prior somatostatin-analog therapy required in patients with midgut carcinoid tumors
* Minimum 4 weeks since completion of prior treatment (investigational or other). Prior treatment with chemotherapy, radiotherapy, hepatic artery embolization, surgery or other therapeutic agents is allowed.
* Treatment related toxicity should have returned to baseline and/or ≤grade 1 prior to study treatment.
* Prior or concurrent therapy with somatostatin analogs is permitted for the control of hormone-mediated symptoms, provided patient has been on a stable dose for at least 2 months and progressive disease on somatostatin analogs (SSTa) has been documented
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Women of childbearing potential must have a negative serum pregnancy test within 14 days prior to treatment.
* Ability to sign informed consent
* Willingness and ability to comply with scheduled visits, laboratory tests and other study procedures

Exclusion Criteria:

* Poorly differentiated, high-grade (e.g. small cell or large cell) neuroendocrine carcinomas are excluded.
* Pancreatic neuroendocrine tumors (NETs), paragangliomas, pheochromocytomas and medullary thyroid cancers are excluded.
* Adenocarcinoid tumors and goblet cell carcinoid tumors are excluded.
* Prior antiangiogenic therapy with a dedicated vascular endothelial growth factor (VEGF) pathway inhibitor
* Clinically apparent central nervous system metastases
* Any of the following within 12 months prior to study: myocardial infarction, uncontrolled angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident, or transient ischemic attack
* Deep venous thrombosis or pulmonary embolism within 6 months of study
* Major surgery 4 weeks prior to enrollment
* Inability to take oral medication or prior surgical procedures affecting absorption (including total gastric resection)
* Active gastrointestinal bleeding, if transfusion dependent
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 28 days
* History of pulmonary hemorrhage or evidence of significant hemoptysis
* History of serious non-healing wound, ulcer, or bone fracture within the past 28 days
* Pre-existing thyroid abnormality allowed provided thyroid function can be controlled with medication.
* Current use or anticipated need for treatment with drugs that are known potent CYP3A4 inhibitors (i.e. grapefruit juice, verapamil, ketoconazole, miconazole, itraconazole, erythromycin, clarithromycin, indinavir, saquinavir, ritonavir, nelfinavir, etc.)
* Current use or anticipated need for treatment with drugs that are known inducers of CYP3AR or CYP1A2 (i.e carbamazepine, dexamethasone, omeprazole, phenobarbital, phenytoin, rifampin, St. John's Wart, etc.)
* Uncontrolled serious medical or psychiatric illness. Patients with a "currently active" second malignancy other than non-melanoma skin cancers, carcinoma in situ of the cervix, resected incidental prostate cancer (staged pathological tumor-2 (pT2) with Gleason Score ≤ 6 and postoperative prostatic specific antigen (PSA) < 0.5 ng/mL), or other adequately treated carcinoma-in-situ are ineligible. Patients are not considered to have a "currently active" malignancy if they have completed therapy and are free of disease for ≥3 years.
* Pregnant or lactating women, or adults of reproductive potential who are not using effective birth-control methods.
* Prior antitumor therapy within 4 weeks of enrollment (with exception of somatostatin analogs)
* Liver-directed therapy within 2 months of enrollment. Prior treatment with radiotherapy (including radio-labeled spheres and/or cyberknife, hepatic arterial embolization (with or without chemotherapy) or cryotherapy/ablation is allowed if these therapies did not affect the areas of measurable disease being used for this protocol or if progressive disease can be documented in the previously treated area.
* Recent infection requiring systemic anti-infective treatment that was completed ≤14 days prior to enrollment (with the exception of uncomplicated urinary tract infection or upper respiratory tract infection)
* Uncontrolled hypertension (blood-pressure >140/90). Patient with baseline hypertension may be eligible after initiation of antihypertensive therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-10-25 (Actual); Primary Completion 2017-01-11 (Actual); Study Completion 2018-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Strosberg, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (2):
- United States (2):
  - University of California San Francisco (UCSF), San Francisco, California
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida and the UCSF Comprehensive Cancer Center, University of California, San Francisco, California, from October 2011 through January 2014.
Groups:
- Axitinib Administration: The investigational drug used in this study is axitinib, and is available as tablets.
Period: Overall Study
Arm/Group | Axitinib Administration
Started | 30
Completed | 22
Not Completed | 8
Not completed — Early withdrawal due to toxicity | 8

BASELINE CHARACTERISTICS:
Population: All participants.
Arm/Group | Axitinib Administration
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 14
Age, Continuous [Median (Full Range); unit: years] | 64 [35 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 13
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Rate of Progression Free Survival (PFS)
Description: Progression-free survival rate at 12 months. PFS: determined as the time from administration of the initial dose of axitinib until objective tumor progression using Response Evaluation Criteria In Solid Tumors (RECIST), or death. Progressive Disease (PD) Appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions. Unequivocal progression should not normally trump target lesion status. It must be representative of overall disease status change, not a single lesion increase. Stable Disease (SD): Neither sufficient shrinkage to qualify for Partial Response (PR) nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: 12 Months
Population: All participants.
Measure: Number; unit: percentage of participants
Arm/Group | Axitinib Administration
Number analyzed (Participants) | 30
percentage of participants | 74.5

2. Primary Outcome: Median Progression Free Survival
Description: Post follow-up progression free survival at time of analysis.
Time Frame: Up to 36 Months
Population: All participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Axitinib Administration
Number analyzed (Participants) | 30
months | 26.7 [11.4 to 35.1]

3. Secondary Outcome: Tumor Response Rate
Description: Tumor response rate using RECIST. Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: 12 Months
Population: All participants evaluable at time of analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Axitinib Administration
Number analyzed (Participants) | 22
Participants
  Partial response | 1
  Stable disease | 21

4. Secondary Outcome: 24 Month Overall Survival (OS) Rate
Description: Overall survival by Kaplan Meier, determined from the time of drug administration to death from any cause. The effect of an intervention is assessed by measuring the number of subjects survived or saved after that intervention over a period of time. The time starting from a defined point to the occurrence of a given event, for example death is called as survival time and the analysis of group data as survival analysis.
Time Frame: 24 months
Population: All participants
Measure: Number; unit: percentage of participants
Arm/Group | Axitinib Administration
Number analyzed (Participants) | 30
percentage of participants | 74.3

5. Secondary Outcome: Time to Treatment Failure
Description: Time to Treatment Failure: Time from administration of the initial dose of axitinib until study discontinuation for any reason (e.g., disease progression, toxicity, death, withdrawal of consent).
Time Frame: 12 Months
Population: All participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Axitinib Administration
Number analyzed (Participants) | 30
months | 9.6 [5.5 to 12]

6. Secondary Outcome: Occurrence of Possibly Related Adverse Events (AEs)
Description: Grade 2 through 4 toxicities considered at least possibly related to treatment. Percentage of participants affected per category. Safety assessments will consist of monitoring and recording all adverse events and serious adverse events, the regular monitoring of hematology and blood chemistry parameters and regular physical examinations. Adverse events will be evaluated continuously throughout the study. Safety and tolerability will be assessed according to the National Institute of Health/National Cancer Institute (NIH/NCI) Common Terminology Criteria for Adverse Events version 4 (CTCAE v4) available at: http://ctep.cancer.gov/protocolDevelopment/electronic_applications/ctc.htm.
Time Frame: 12 Months
Population: All participants.
Measure: Number; unit: percentage of participants
Arm/Group | Axitinib Administration
Number analyzed (Participants) | 30
percentage of participants
  Hypertension | 87
  Abdominal pain | 17
  Diarrhea | 17
  Nausea | 13
  Vomiting | 7
  Mucositis | 3
  Oral pain | 3
  Headache | 20
  Confusion | 3
  Insomnia | 3
  Syncope | 3
  Anxiety | 3
  Intracranial hemorrhage | 3
  Fatigue | 27
  Weight loss | 6
  Anorexia | 3
  Myalgia | 3
  Dehydration | 10
  Hypothyroidism | 3
  Increased transaminases | 3
  Increased alkaline phosphatase | 10
  Increased gamma-glutamyl transferase | 3
  Urinary tract infection | 3
  Right ventricular dysfunction | 3
  Pain in extremity | 3
  Hand-foot syndrome | 2

ADVERSE EVENTS:
Time Frame: 3 years, 10 months
Arm/Group | Axitinib Administration
Serious Adverse Events (participants affected / at risk) | 12/30
Other Adverse Events (participants affected / at risk) | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Axitinib Administration (N=30)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Aortic valve disease (Cardiac disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Colitis (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Pancreatitis (Gastrointestinal disorders) | 2 (3)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1)
Rectal ulcer (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Chills (General disorders) | 1 (3)
Fatigue (General disorders) | 3 (3)
Fever (General disorders) | 1 (3)
Bile duct stenosis (Hepatobiliary disorders) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Intracranial hemorrhage (Nervous system disorders) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1)
Nervous system disorders - Other, neurologic changes (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Hypertension (Vascular disorders) | 2 (2)
Hypotension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Axitinib Administration (N=30)
Anemia (Blood and lymphatic system disorders) | 7 (7)
Hypothyroidism (Endocrine disorders) | 3 (3)
Dry eye (Eye disorders) | 2 (3)
Abdominal pain (Gastrointestinal disorders) | 8 (16)
Anal mucositis (Gastrointestinal disorders) | 2 (6)
Anal pain (Gastrointestinal disorders) | 2 (3)
Bloating (Gastrointestinal disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 7 (19)
Diarrhea (Gastrointestinal disorders) | 12 (27)
Dry mouth (Gastrointestinal disorders) | 4 (4)
Dyspepsia (Gastrointestinal disorders) | 3 (4)
Flatulence (Gastrointestinal disorders) | 3 (4)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 3 (5)
Hemorrhoids (Gastrointestinal disorders) | 5 (7)
Mucositis oral (Gastrointestinal disorders) | 5 (7)
Nausea (Gastrointestinal disorders) | 12 (19)
Oral pain (Gastrointestinal disorders) | 3 (6)
Rectal hemorrhage (Gastrointestinal disorders) | 2 (2)
Rectal pain (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 6 (8)
Edema limbs (General disorders) | 3 (4)
Fatigue (General disorders) | 17 (32)
General disorders and administration site conditions - Other, specify (General disorders) | 3 (7)
Non-cardiac chest pain (General disorders) | 2 (3)
Pain (General disorders) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (3)
Alanine aminotransferase increased (Investigations) | 4 (5)
Alkaline phosphatase increased (Investigations) | 4 (8)
Blood bilirubin increased (Investigations) | 3 (5)
Creatinine increased (Investigations) | 4 (4)
Platelet count decreased (Investigations) | 8 (18)
Weight loss (Investigations) | 10 (10)
Anorexia (Metabolism and nutrition disorders) | 9 (9)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 10 (22)
Hyperkalemia (Metabolism and nutrition disorders) | 4 (8)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (5)
Hypoglycemia (Metabolism and nutrition disorders) | 3 (6)
Hypokalemia (Metabolism and nutrition disorders) | 4 (6)
Hyponatremia (Metabolism and nutrition disorders) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (10)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (4)
Dizziness (Nervous system disorders) | 5 (7)
Headache (Nervous system disorders) | 14 (21)
Paresthesia (Nervous system disorders) | 2 (2)
Anxiety (Psychiatric disorders) | 4 (4)
Confusion (Psychiatric disorders) | 2 (3)
Depression (Psychiatric disorders) | 4 (4)
Insomnia (Psychiatric disorders) | 7 (11)
Proteinuria (Renal and urinary disorders) | 4 (7)
Renal and urinary disorders - Other (Renal and urinary disorders) | 2 (3)
Reproductive system and breast disorders - Other (Reproductive system and breast disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 10 (12)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 5 (6)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 3 (4)
Hematoma (Vascular disorders) | 2 (3)
Hypertension (Vascular disorders) | 26 (266)

LIMITATIONS AND CAVEATS:
Results are limited by a relatively high rate of participant withdrawal before progression due to toxicity. Post analysis, 2 participants are still on study at UCSF.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes